CLINICAL TRIAL: NCT01998165
Title: An Open-Label Study to Evaluate the Efficacy and Safety of JNJ-268229 in Pediatric Subjects General Anesthetised
Brief Title: A Study to Evaluate the Safety and Efficacy of Ultiva (Remifentanil Hydrochloride) in Pediatric Participants General Anesthetised
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR102524; ULTIVAANS3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-11-15; First posted 2013-11-28 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Anesthesia
Keywords: Anesthesia; Remifentanil; Ultiva
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remifentanil (0.25 µg/kg/min) (Experimental)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — After intubation, continuous intravenous infusion of remifentanil (0.25 µg/kg/min) is started, while anesthesia is maintained with inhaled or intravenous anesthetics. In cases where sedation by general anesthetics and analgesia by lidocaine does not seem to provide a sufficient means of analgesia at the time of intubation, remifentanil may be used, beginning before intubation. The rate of infusion may be adjusted while monitoring the subject's general condition in 25% to 100% increments or in 25% to 50% decrements every 2 to 5 minutes, but should not exceed 1.3 µg/kg/min.
  Other Names: remifentanil hydrochloride (JNJ-268229)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JNJ-268229 (Ultiva /Remifentanil Hydrochloride) in pediatric participants between 1 and 15 years of age during maintenance of general anesthesia.

DETAILED DESCRIPTION:
This is multicenter, open-label (identity of assigned study drug will be known) one-arm study in pediatric participants receiving general anesthesia. The participants are children aged 1-15 years old, planned to undergo head and neck, thoracic (except heart), urological, orthopedic or plastic surgery. Approximately 80 participants will be enrolled in this study. These participants are divided into two groups by age (1-6 and 7-15 years old). Pharmacokinetic (what the body does to the drug,) blood samples will be collected from at least 3 participants between the ages of 1 and 6 years and at least 3 participants between the ages of 7 and 15 years from 15 minutes after the start of infusion to the end of infusion of the study drug . The study consists of 4 phases: screening phase, treatment phase, recovery phase and follow-up phase. Screening for eligible participants will be performed within 14 days before administration of the study drug. The safety and tolerability of study drug will be evaluated by physical examinations, electrocardiogram (ECG), clinical laboratory tests, vital signs, and adverse events (AEs) according to the Time and Events Schedule. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants scheduled to receive surgery under general anesthesia, necessitating airway securing with tracheal intubation and analgesia with opioid analgesics
* American Society of Anesthesiologists (ASA) Physical Status Classification is I or II at the time of operation planning
* Participants scheduled to receive operations estimated to take 30 minutes or more from skin incision i.e. Head and neck, thoracic (except heart), intraperitoneal, ophthalmological, otorhinolaryngological, urological, orthopedic or plastic surgery
* Girls having undergone menarche are eligible only if the urine pregnancy test at the time of screening is negative Exclusion Criteria:-
* Chronic use of opioid analgesics or their use within 12 hours before the planned start of general anesthesia - Hypersensitivity to opioid analgesics or local anesthetics
* History of jaundice or unexplained fever induced by halogenated anesthetics
* Unstable hemodynamics (eg. congenital heart disease, congenital diaphragmatic hernia) Ideal body weight is not within the 10th to 90th percentile received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned first dose of study drug or is currently enrolled in an investigational study

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with positive response to skin incision | 5-minute assessment period after skin incision
  Positive response is defined by the presence of at least one of below listed conditions: Heart rate increased >20% above baseline (that is measured under stable hemodynamics after intubation, and 1-5 minutes before the planned start of skin incision) for >1 minute); Systolic blood pressure increased >20% above baseline (that is measured under stable hemodynamics after intubation, and 1-5 minutes before the planned start of skin incision) for >1 minute; Gross movement, swallowing, eye opening (if there are patches on the eyes, this assessment might be not evaluated) or grimacing and sweating, lachrymation or mydriasis.

SECONDARY OUTCOMES:
Hemodynamics stability | 5-60 minutes before the start of intubation, 1-5 minutes before the planned start of the first skin incision. and 240 minutes after completion of anesthesia or skin closure
  Heart Rate and Blood Pressure increased >20% above baseline that is measured under stable hemodynamics after intubation, and 1-5 minutes before the planned start of skin incision for less than or equal to 1 minute.
Drugs used to deal with insufficient anesthesia (inadequate anesthesia) or excessive anesthesia | Time interval between completion of anesthesia and extubation
  The time interval between completion of anesthesia and extubation is calculated based on both the time upon completion of general anesthesia and the time upon completion of extubation and recorded.
Assessment on analgesic effect | 240 minutes after completion of anesthesia
  Assess an analgesic effect of JNJ-268229 during operation on 3-point ranging from "effective / not effective / undeterminable" generally.
Total dose level of remifentanil | 1-5 minutes before the planned start of the first skin incision. and 240 minutes after completion of anesthesia or skin closure
  The overall use (including dose increase/decrease, time of dose increase/decrease and start time of single supplemental bolus injection, etc) of remifentanil will be recorded.
Total concomitant anesthetic dose level | 1-5 minutes before the planned start of the first skin incision. and 240 minutes after completion of anesthesia or skin closure
  The overall use (drug name, dose and start time, etc) of the inhaled or intravenous anesthetics used for general anesthesia
Time from completion of anesthesia to resumption of spontaneous respiration | 1-5 minutes before the planned start of the first skin incision. and 240 minutes after completion of anesthesia or skin closure
  The time taken from completion of anesthesia to resumption of spontaneous respiration is calculated based on both the time upon completion of general anesthesia and the time upon confirmation of resumed spontaneous respiration and recorded.
Time until arrival of Steward Postanesthetic Recovery Score at 6 | 240 minutes after completion of anesthesia or skin closure
  Recovery Score is rated as Consciousness,Airway and Movement
Time from completion of anesthesia to discharge from the recovery room | 240 minutes after completion of anesthesia or skin closure
  Anesthesia is calculated based on both the time upon completion of general anesthesia and the time upon discharge from the operating /recovery room.
Respiratory stability | 5-60 minutes before the start of intubation, 1-5 minutes before the planned start of the first skin incision. and 240 minutes after completion of anesthesia or skin closure
  Heart Rate and Blood Pressure increased >20% above baseline that is measured under stable hemodynamics after intubation, and 1-5 minutes before the planned start of skin incision for less than or equal to 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (9):
- Japan (9):
  - Asahikawa
  - Kobe
  - Kure
  - Kurume
  - Ohmura
  - Osaka
  - Shimajiri
  - Shimotsuke
  - Tokyo

REFERENCES:
- See also: An Open-Label Study to Evaluate the Efficacy and Safety of JNJ-268229 in Pediatric Subjects General Anesthetised — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=5192&filename=CR102524_CSR.pdf